CLINICAL TRIAL: NCT05171504
Title: Detection of Lactoferrin and Iron in Seminal Plasma and Their Possible Relation to Fertility Status in Varicocele: A Case-control Study
Brief Title: Lactoferrin and Iron in Seminal Plasma of Varicocele
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marilyn Sameh, Principle investigator, Assiut University
Other Study IDs: lactoferrin,iron in varicocele
Record Dates: First submitted 2021-10-16; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Varicocele
Keywords: lactoferrin, iron
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — semen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- I , Infertile males with varicocele: Lactoferrin , iron in seminal plasma and semen analysis from Infertile patients with varicocele
- II , infertile males due to other causes than varicocele: Lactoferrin , iron in seminal plasma and semen analysis from infertile patients due to other causes than varicocele
- III , fertile males: Lactoferrin , iron in seminal plasma and semen analysis from fertile males with history of childbirth within the previous year

SUMMARY:
Infertility is defined by World Health Organization (WHO) as a disease of reproductive system characterized by failure to achieve clinical pregnancy even after 12 months or more of regular unprotected sexual intercourse. It affects around 15% of all couples, that is 48.5 million couples worldwide.

Male infertility has emerged as an important cause of infertility worldwide. There are many factors affecting male fertility and research is going on to know impact of various factors on sperm functions.Male infertility affects 30:40% of cases.

Infertility could be due to different aetiologies. Among the possible causes are genetic factors, obstructive disorders (congenital absence of vas deferens), varicocele and testicular dysgenesis. However, some cases of male infertility are idiopathic.

DETAILED DESCRIPTION:
Varicocele is considered as the second most common cause of infertility. In the general population, approximately 15% of adult men have varicocele, but in the population of infertile men, the prevalence rises to 40% of cases with primary infertility and 80% in secondary infertility .

Varicocele is characterised by dilated veins of the pampiniform plexus which are responsible for the testicular blood drainage.Varicocele can affect fertility through hypoxia of the testicular tissues, germ cell apoptosis, oxidative stress, reflux of toxic metabolites from the renal/adrenal tissues and hyperthermia of the testis.

Semen analysis is the gold standard diagnostic test for male infertility. Seminal plasma is considered a gold mine for male fertility as it contains molecules from male reproductive glands which play important role in sperm function.

Lactoferrin is an iron-binding globular glycoprotein that act as immunomodulator mainly at mucosal level. In general, lactoferrin plays important role in the regulation of iron absorption, the modulation of immune responses, and has anti-microbial, anti-viral, antioxidant, anticancer, and anti-inflammatory activities.

Lactoferrin is found in various exocrine fluids and blood plasma. It is secreted from the prostate and seminal vesicles in humans. The physiological role of the lactoferrin in the male reproductive tract remains unclear.

Few studies have investigated the effect of lactoferrin on semen quality in humans. A recent study has demonstrated that lactoferrin expression on cells of seminal fluid was associated with worse sperm concentration and morphology, considering it as a possible novel marker of male infertility. Other studies showed that seminal lactoferrin concentrations were raised in patient groups with oligozoospermia and oligoasthenozoospermia.

Iron is an essential trace nutrient that plays an important role in general health and fertility. It is not essentially toxic, but disturbances can appear due to prolonged intake of high doses or dysfunction in the regulatory mechanism.

Iron is one of the trace elements that present in semen.It participates in oxygenation and reduction processes, entering into the composition of many enzymes and metalloprotein compounds. It has been reported that iron can cause an increase in sperm damage.

The toxicity of iron could result from the formation of hydroxyl free radicals. Iron-induced oxidative stress may induce lipid peroxidation, which has been shown to result in deterioration of sperm morphology and motility. So, iron is highly toxic if accumulated in large quantities. Also,the excess or deficiency may lead to defective spermatogenesis and to fertility impairment.

Most of the previous researches on the effect of iron on sperm function have shown increased level of seminal iron in sub-fertile than fertile men. In addition, significant higher concentrations of seminal iron were detected in asthenozoospermic and teratozoospermic groups.

On the contrary, a study has demonstrated that iron level and other trace elements were significantly lower in seminal fluid of asthenozoospermic subjects in comparison with normozoospermic men. In that study, although higher levels of iron were detected in men with normal semen analysis, these higher levels adversely affected sperm motility in this group.

ELIGIBILITY:
Inclusion Criteria:

* Group I will include infertile patients with varicocele that is diagnosed clinically and by doppler scrotal ultrasonography.
* Group II will include infertile patients due to other causes than varicocele
* Group III will include fertile men with history of childbirth within the previous year.

Exclusion Criteria:

The patients will be excluded from the group I in the following conditions:

1. History or evidence of Genital tract infection.
2. History or evidence of hormonal/chromosomal abnormalities.
3. History or evidence of chronic debilitating diseases.
4. History of hormonal treatment or chemotherapy.
5. Low semen volume less than 1.5 ml.
6. Severe oligozoospermia less than 5x10*6 /ml.
7. Azoospermia.

Ages: 20 Years to 50 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes
Study Population: The participants will be divided in to three equal groups:
  Group I: will include 25 patients with varicocele seeking medical advice for infertility.
  Group II: will include 25 patients seeking medical advice for infertility due to other causes than varicocele as a control group.
  Group III: will include 25 fertile male participants as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Detection of lactoferrin and iron in seminal plasma and their possible relation to fertility status in varicocele | 6 months
  Correlation of the level of lactoferrin and iron in seminal plasma with semen parameters in infertile patients with varicocele , infertile patients due to other causes than varicocele and fertile men.
  Evaluation the level of lactoferrin in seminal plasma by using ELISA method and the level of iron in seminal plasma by semiautomated colorimetric method.

REFERENCES:
- [Background] Collodel G, Signorini C, Nerucci F, Gambera L, Iacoponi F, Moretti E. Semen Biochemical Components in Varicocele, Leukocytospermia, and Idiopathic Infertility. Reprod Sci. 2021 Jan;28(1):91-101. doi: 10.1007/s43032-020-00260-0. Epub 2020 Jul 22. PMID 32696238
- [Background] Aydemir B, Kiziler AR, Onaran I, Alici B, Ozkara H, Akyolcu MC. Impact of Cu and Fe concentrations on oxidative damage in male infertility. Biol Trace Elem Res. 2006 Sep;112(3):193-203. doi: 10.1385/BTER:112:3:193. PMID 17057258
- [Background] Kamal HM, El-Fallah AA, Abdelbaki SA, Khalil MM, Kamal MM, Behiry EG. Association between seminal granulysin and malondialdehyde in infertile men with varicocele and the potential effect of varicocelectomy. Andrologia. 2020 Jul;52(6):e13579. doi: 10.1111/and.13579. Epub 2020 Apr 9. PMID 32271478
- [Background] Kasperczyk A, Dobrakowski M, Czuba ZP, Kapka-Skrzypczak L, Kasperczyk S. Influence of iron on sperm motility and selected oxidative stress parameters in fertile males - a pilot study. Ann Agric Environ Med. 2016 Jun 2;23(2):292-6. doi: 10.5604/12321966.1203893. PMID 27294635
- [Background] Hao L, Shan Q, Wei J, Ma F, Sun P. Lactoferrin: Major Physiological Functions and Applications. Curr Protein Pept Sci. 2019;20(2):139-144. doi: 10.2174/1389203719666180514150921. PMID 29756573
- [Background] Buckett WM, Luckas MJ, Gazvani MR, Aird IA, Lewis-Jones DI. Seminal plasma lactoferrin concentrations in normal and abnormal semen samples. J Androl. 1997 May-Jun;18(3):302-4. PMID 9203059
- [Background] Ammar O, Houas Z, Mehdi M. The association between iron, calcium, and oxidative stress in seminal plasma and sperm quality. Environ Sci Pollut Res Int. 2019 May;26(14):14097-14105. doi: 10.1007/s11356-019-04575-7. Epub 2019 Mar 9. PMID 30852746
- [Background] Marzec-Wroblewska U, Kaminski P, Lakota P, Szymanski M, Wasilow K, Ludwikowski G, Kuligowska-Prusinska M, Odrowaz-Sypniewska G, Stuczynski T, Michalkiewicz J. Zinc and iron concentration and SOD activity in human semen and seminal plasma. Biol Trace Elem Res. 2011 Oct;143(1):167-77. doi: 10.1007/s12011-010-8868-x. Epub 2010 Oct 6. PMID 20924714
- [Background] Kikuchi M, Takao Y, Tokuda N, Ohnami Y, Orino K, Watanabe K. Relationship between seminal plasma lactoferrin and gonadal function in horses. J Vet Med Sci. 2003 Nov;65(11):1273-4. doi: 10.1292/jvms.65.1273. PMID 14665762
- [Background] Gill K, Kups M, Harasny P, Machalowski T, Grabowska M, Lukaszuk M, Matuszewski M, Duchnik E, Fraczek M, Kurpisz M, Piasecka M. The Negative Impact of Varicocele on Basic Semen Parameters, Sperm Nuclear DNA Dispersion and Oxidation-Reduction Potential in Semen. Int J Environ Res Public Health. 2021 Jun 2;18(11):5977. doi: 10.3390/ijerph18115977. PMID 34199549
- [Background] Hashemi MM, Behnampour N, Nejabat M, Tabandeh A, Ghazi-Moghaddam B, Joshaghani HR. Impact of Seminal Plasma Trace Elements on Human Sperm Motility Parameters. Rom J Intern Med. 2018 Mar 1;56(1):15-20. doi: 10.1515/rjim-2017-0034. PMID 28865234
- [Background] Kumar N, Singh NK. "Emerging role of Novel Seminal Plasma Bio-markers in Male Infertility: A Review". Eur J Obstet Gynecol Reprod Biol. 2020 Oct;253:170-179. doi: 10.1016/j.ejogrb.2020.08.015. Epub 2020 Aug 24. PMID 32871440
- [Background] Omes C, De Amici M, Tomasoni V, Todaro F, Torre C, Nappi RE. Myeloperoxidase and lactoferrin expression in semen fluid: Novel markers of male infertility risk? Immunobiology. 2020 Sep;225(5):151999. doi: 10.1016/j.imbio.2020.151999. Epub 2020 Aug 5. PMID 32962819